CLINICAL TRIAL: NCT00114270
Title: Evaluating the Effect of Letrozole With or Without Concomitant Zoledronic Acid on Estrogen Responsive Targets in Postmenopausal Women
Brief Title: Letrozole With or Without Zoledronate in Treating Healthy Postmenopausal Women With High Breast Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000430927; UVACC-HIC-11019; UVACC-31003
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2006-04

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: breast cancer; osteoporosis
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Letrozole; Zoledronic Acid

INTERVENTIONS:
Drug: letrozole
Drug: zoledronic acid

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may prevent breast cancer by lowering the amount of estrogen the body makes. Zoledronate may prevent bone loss caused by letrozole. Giving letrozole together with zoledronate may prevent breast cancer and reduce bone loss.

PURPOSE: This randomized clinical trial is studying letrozole and zoledronate to see how well they work compared to letrozole and placebo or placebo alone in treating healthy postmenopausal women with high breast density.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the percent change in breast density in healthy postmenopausal women with high breast density treated with placebo only vs letrozole and placebo vs letrozole and zoledronate.
* Compare the percent change in biochemical markers of bone turnover in participants treated with these regimens.

Secondary

* Compare the bone density in participants treated with these regimens.
* Compare growth hormone release and insulin-like growth factor levels in participants treated with these regimens.
* Compare the incidence and severity of adverse events in participants treated with these regimens.

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter, pilot study. Participants are stratified according to prior hormone replacement therapy (HRT) use (discontinued HRT > 5 years ago or no prior HRT use vs discontinued HRT 1-5 years ago). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Participants receive oral placebo once daily for 12 months and placebo IV over 15 minutes on day 0 and at 6 months.
* Arm II: Participants receive oral letrozole once daily for 12 months and placebo IV over 15 minutes on day 0 and at 6 months.
* Arm III: Participants receive oral letrozole once daily for 12 months and zoledronate IV over 15 minutes on day 0 and at 6 months.

In all arms, treatment continues in the absence of unacceptable toxicity.

After completion of study treatment, participants are followed at 3 months.

PROJECTED ACCRUAL: A total of 120 participants (40 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participant
* Postmenopausal for > 5 years
* Breast density ≥ 50% by digitized mammography
* No history of breast cancer, breast implant, or gynecological malignancy
* No osteoporosis or postmenopausal fractures

  * T-scores ≥ -2.0 by dual-energy x-ray absorptiometry (DEXA) scan

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* See Disease Characteristics

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* AST or ALT ≤ 3 times normal

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* No cardiac disease

Other

* Nonsmoker
* Vitamin D ≥ 15 ng/mL
* No history of chronic medical or psychiatric condition or laboratory abnormality that would preclude study compliance or participation
* No alcohol consumption of > 2 alcoholic drinks per day
* No malabsorption

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* At least 1 year since prior hormone replacement therapy
* No concurrent steroids, parathyroid hormone, or raloxifene

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No other concurrent medication known to affect calcium and bone metabolism (e.g., anticoagulants, antiseizure medications, bisphosphonates, or calcitonin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2004-05; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ailleen Heras-Herzig, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States